CLINICAL TRIAL: NCT01420939
Title: Biomarkers-Driven Development of Experimental Therapeutics for Traumatic Brain Injury
Brief Title: Developing Therapies for Traumatic Brain Injury
Status: Terminated | Type: Observational
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110213; 11-NR-0213
Record Dates: First submitted 2011-08-19; First posted 2011-08-22 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2013-05-21

CONDITIONS: Traumatic Brain Injury
Keywords: TBI; Brain; Traumatic Brain Injury; Biomarkers; Healthy Volunteer; HV
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- A person who has a traumatic brain injury (TBI) -- also called concussion -- can have serious and long-lasting effects. Doctors who treat TBI need more information about how the brain changes over time in people with TBI and how well a person recovers from it. To make existing TBI treatments more effective and develop new ones, researchers want to look more closely at how TBI affects people both physically and psychologically.

Objectives:

- To collect medical information from people with recent traumatic brain injury and compare this information to that of healthy volunteers and of persons who have had injuries to other parts of their bodies besides their heads (such as broken bones, orthopedic injuries, after surgery).

Eligibility:

3 groups of people between the ages of 18 and 70 years will be asked to take part.

* Persons who have had a traumatic brain injury (or concussion ) within the past 30 days, OR
* Persons who are healthy and have never had a traumatic brain injury, OR
* Persons who have had an injury within the past 30 days to a part of their body other than the head (such as a broken bone, orthopedic injury, surgery)

Design:

* This study requires two outpatient visits each lasting 1 1/2 days. The 2 visits will be about 30 days apart. Persons with TBI and non-TBI injuries must have their first visit within 30 days of their injury.
* Screening: Participants will be screened with a medical history, physical examination, blood tests and electrocradiogram (ECG a routine heart test).
* The research will involve:

  1. Giving blood samples (no more than 75 ml each visit).
  2. Having tests of memory, attention, concentration, and thinking (neuropsychological testing).
  3. Having imaging studies of the head including magnetic resonance imaging (MRI) and positron emission tomography (PET) scans.
* Persons with TBI will have the same tests at Visit 1 and 2. Healthy controls and persons with non-TBI injuries will have the same tests at Visit 1 as listed above. But, at Visit 2, they will not have brain MRIs or PETs.
* No treatments will be provided as part of this research protocol.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is the leading cause of death and disability in people under age 45 in industrialized countries, but there is no specific treatment available for TBI. Circulating endothelial progenitor cells (EPC) are markers of vascular injury that are mobilized after signaling with cytokines, interleukins, MMP9 and other biomarkers (BM) that may be detected in blood. However, the relation of EPC and these BM to TBI severity has not been quantified. MRI measurements of lesion volume provide an objective method for TBI severity assessment and outcome prediction. Moreover, diffusion tensor imaging (DTI) is sensitive to detect TBI-related axonal injury, and PET (positron emission tomography) is useful in functional interpretation of image findings. This cross-sectional study aims to determine whether EPC and other BM are associated with MRI, DTI and PET findings, and with functional outcomes in TBI patients.

OBJECTIVES:

The primary objective of the study is to evaluate levels of EPC and other BMs participating in EPC mobilization in TBI patients in comparison to the healthy volunteers and to the non-TBI trauma controls. The second objective is to relate EPC and BM levels to TBI severity quantified by functional and radiological evaluations (MRI, DTI and PET). The third objective is to determine, if there is a relationship between the level of EPC and other BM and functional outcomes.

POPULATION:

100 male or female participants between 18 and 70 years of age will be enrolled within 30 days of a moderate TBI (classified as Glasgow Coma Scale (GCS) of 9-12) or mild TBI (GCS 13-15). If participants had post-traumatic amnesia (PTA) it must have lasted less than 7 days and any loss of consciousness (LOC) must have lasted less than 24 hours. Fifty healthy volunteers and 50 persons with non-TBI injuries (such as broken bones, orthopedic injuries or surgery) will be enrolled.

RESEARCH DESIGN:

Before participating in this protocol, TBI and non-TBI injured participants must have received routine clinical evaluations for their injuries in hospitals, doctors offices or other medical facilities. They may be referred to the NIH Clinical Center after discharge or they may be self-referred. They must be willing to have their medical records sent to the NIH to assure that their injuries fit the protocol inclusion criteria. Healthy volunteers may be recruited from families of other participants but most will be recruited through the NIH Patient Recruitment and Public Liaison Office (PRPL).

This is an outpatient, observational study. Eligible participants will come to the NIH for two 1 1/2 day outpatient visits separated by 30 days. Persons with TBI will have the same tests at each of their two visits: a history and physical exam, electrocardiogram, research blood draws (no more than 75 ml each visit), pregnancy and HIV testing, neuropsychological testing, head magnetic resonance imaging (MRI) scan, and positron emission tomography scan (PET scan). Healthy controls and persons with non-TBI injuries will have the same tests at visit 1 as listed above. At visit 2, they will have all the same tests except they will not have brain MRIs or PETs.

IMPORTANCE:

This study will provide novel data regarding the association of levels of EPC and the blood BMs with severity of imaging-positive TBI. This study will provide a foundation for the development of interventional trials aiming to improve neovascularization in TBI patients.

ELIGIBILITY:
* INCLUSION CRITERIA FOR TBI PATIENTS:

To be included, TBI patients must meet all of the following criteria:

* Between 18 and 70 years of age
* Had head injury within the previous 30 days.
* Had a moderate TBI classified as GCS 9-12 or a mild TBI classified as GCS 13-15 at the first ER or other medical examination. If LOC existed, it may not have lasted more than 24 hours. If PTA existed it may not be more than 7 days.
* Admitted to an inpatient unit, ED, and/or evaluated in a doctors' office because of head trauma.
* Injury occurred less than 30 (plus 5) days before enrollment
* Willingness to provide permission to allow release of medical records related to these injuries.

INCLUSION CRITERIA FOR HEALTHY VOLUNTEERS:

Healthy volunteers will be eligible for enrollment if they meet the following inclusion requirements:

* Between 18 and 70 years of age
* Determined to be healthy at the time of screening
* No known previous TBI, even mild (characterized as GCS >13, PTA < 1 day LOC < 30 min)

INCLUSION CRITERIA FOR NON-TBI TRAUMA CONTROLS:

Non-TBI trauma controls will be eligible for enrollment if they meet the following criteria:

* Between 18 and 70 years of age
* Evaluated in an emergency department or in a physician s office or admitted to an inpatient unit because of isolated traumatic injury resulting in a fracture (e.g, limbs, ribs) or other orthopedic injury (ligament, tendon or joint injury) or non-life threatening condition requiring surgery (appendectomy, etc.).
* No known previous TBI, even mild (characterized as GCS > 13, PTA < 1 day LOC < 30 min)
* Evaluated within 30 (plus 5) days after the trauma
* Willingness to provide permission to allow release of medical records related to these injuries.

EXCLUSION CRITERIA FOR ALL STUDY PARTICIPANTS:

Study participants will be excluded from the study if he/she has one or more of the following:

* Are not able to read and understand English to complete outcome assessments and neurological scales
* Progressive or unstable disease of any body system including cardiovascular, pulmonary, gastrointestinal, central nervous system, psychiatric, endocrine, hematologic, renal, or immunologic disorders
* Alcohol dependence/substance abuse history within the past 5 years
* Known acute and chronic inflammatory disease (i.e. rheumatoid arthritis, systemic lupus erythematosus, hepatitis, cirrhosis, sepsis, severe periodontosis or HIV infection or AIDS.
* Clinically significant abnormal ECG, or acute myocardial infarction within last 3 months
* Ischemic or hemorrhagic stroke within last 3 months
* History of diabetes
* Currently undergoing evaluation or treatment for chronic illness or presenting with symptoms suggestive of undiagnosed disorders
* Pregnant or lactating women

EXCLUSION CRITERIA FOR BRAIN MRI:

Of the participants and volunteers enrolled under the listed inclusion/exclusion, the following will not be eligible for MRI scanning but will undergo all other study procedures:

* Contraindication to MRI scanning, including certain metal implants or any other device such as: cardiac pacemaker, insulin infusion pump, implanted drug infusion device, cochlear, otologic, or ear implant, transdermal medication patch (nitroglycerine), any metallic implants or objects, body piercing(s), bone/joint pin, screw, nail, plate, wire sutures or surgical staples, shunts, cerebral aneurysms clips, shrapnel or other metal imbedded in a participant s body (such as from war wounds or accidents or previous work in metal fields or machines that may have left any metallic fragments in or near the participant s eyes)
* Previous trauma or accidents in the past with non-certainty that metal objects are still present in the body
* A condition precluding entry into the scanner (e.g. morbid obesity or claustrophobia)
* Pregnant women or women who are breast-feeding.
* Inability to lie flat on back for up to 90 minutes

EXCLUSION CRITERIA FOR BRAIN PET:

* A condition precluding entry into the scanner (e.g. morbid obesity or claustrophobia)
* Pregnancy or breast-feeding
* Blood glucose over 200 mg/dL when measured before the PET scanning
* Previous radiation exposure where the additional exposure from the PET scan would exceed NIH annual limits

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-07-21; Study Completion 2013-05-21

PRIMARY OUTCOMES:
Difference in levels BMs of neovascularization, neuroinflammation, and BM of severity of TBI and epigenetic changes in TBI group in comparison to volunteer group and trauma patients.

SECONDARY OUTCOMES:
Correlation of levels of the BMs of neovascularization, neuroinflammation and severity of TBI to TBI severity assessed by functional outcomes and imaging (MRI, PET) evaluations in TBI patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Gill, Ph.D., Principal Investigator — National Institute of Nursing Research (NINR)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kraus MF, Smith GS, Butters M, Donnell AJ, Dixon E, Yilong C, Marion D. Effects of the dopaminergic agent and NMDA receptor antagonist amantadine on cognitive function, cerebral glucose metabolism and D2 receptor availability in chronic traumatic brain injury: a study using positron emission tomography (PET). Brain Inj. 2005 Jul;19(7):471-9. doi: 10.1080/02699050400025059. PMID 16134735
- [Background] Langlois JA, Rutland-Brown W, Wald MM. The epidemiology and impact of traumatic brain injury: a brief overview. J Head Trauma Rehabil. 2006 Sep-Oct;21(5):375-8. doi: 10.1097/00001199-200609000-00001. PMID 16983222
- [Background] Rutland-Brown W, Langlois JA, Thomas KE, Xi YL. Incidence of traumatic brain injury in the United States, 2003. J Head Trauma Rehabil. 2006 Nov-Dec;21(6):544-8. doi: 10.1097/00001199-200611000-00009. PMID 17122685